CLINICAL TRIAL: NCT04414644
Title: Randomized Study of Daytime vs. Delayed Eating: Effect on Weight and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kelly Allison, Director, Center for Weight and Eating Disorders, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 820064; R21DK100787 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Metabolism; Eating; Circadian Rhythms
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized within subjects, cross-over design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daytime Eating Condition (Experimental): Participants will be asked to eat all of their meals and snacks, as provided by the study, between 0800 and 1900.
  Interventions: Behavioral: Eating Condition
- Delayed Eating Condition (Experimental): Participants will be asked to eat all of their meals and snacks, as provided by the study, between 1200 and 2300.
  Interventions: Behavioral: Eating Condition

INTERVENTIONS:
Behavioral: Eating Condition — Participants will be randomly assigned to eat per the prescribed eating condition for 8 weeks during eating condition 1. They will complete the alternate eating condition for 8 weeks during eating condition 2.

SUMMARY:
The purpose of this study is to determine if, controlling for eating and sleep timing, caloric intake, and exercise, daytime vs. delayed eating affects body mass, adiposity, and energy metabolism in healthy adults.

DETAILED DESCRIPTION:
The study consists of 4 phases - screening & baseline assessment, eating condition 1, wash-out period, and eating condition 2. Before and after each phase participants will complete a 28-hour inpatient assessment at the Clinical and Translational Research Center (CTRC) of the Hospital of the University of Pennsylvania to study the impact of one's eating on body weight and fat content, metabolism, and certain markers of metabolism in the blood.

Screening In order to participate in this study the participants must undergo a complete physical examination and tests of blood and urine. These tests will determine if participants have any conditions that would prevent them from participating in the study, including diabetes or any serious uncontrolled medical condition that may interfere with their participation in the study. Other conditions that would prevent them from taking part are pregnancy or nursing, a sleep disorder, the use of certain medications, or night-shift work. A urine pregnancy test will be given to women at this screening visit.

Participants will also complete several surveys of a psychological nature and participate in a clinical interview. Sleep and exercise schedules are important and will be reviewed during their visits to see if they match with the study requirements. During the 10 days of the screening assessment, participants will keep a log in which they will record all food and beverages that they consume. They will also use these logs to record when they sleep and exercise. Their activity will be measured by a small electronic wrist activity recorder, called an Actigraph (about the size of a wrist watch), during this time. This recorder, similar to a pedometer, records all activity from the arm, and is very useful in determining if and when they get up at night. Study staff will explain how to keep this information during the baseline visit. They will return the activity recorder and log to Dr. Allison for analysis at the end of the 10-days. They are expected to return all study materials, including the Actigraph, log, and questionnaires.

Assessments Following successful completion of the screening period, they will complete the first of four assessment visits. This visit will include 28 hours (overnight) spent at the CTRC, where their meals and snacks will be provided.

They will arrive at the CTRC at the Hospital of the University of Pennsylvania at 7 am. Starting at 8 am, their blood will be drawn every four hours. A thin needle (an introducer) will be inserted into a vein in their forearm, much like an IV line. Very small blood samples, 10 mL (2 teaspoonfuls), will be collected every four hours from 8:00 am on Day 1 through 8:00 am on Day 2. From this blood study staff will measure hormones related to metabolism, sleep, and stress. They will be provided meals and snacks during this time, and they are free to watch television or use their computer or participate in other sedentary pastimes while they are there.

After the blood draws end at 8 am on the second morning, their metabolic rate will be measured. Participants will be asked to fast for 10 hours overnight (they will not be able to eat or drink anything except water for 10 hours starting at 10 pm the night before). Then study staff will measure their resting metabolic rate for 20 minutes. During the measurements, they will lay on their back in bed with a plastic hood/canopy over their head and neck. They will lay still and breathe normally while the air they inhale and exhale is collected in the canopy/hood and analyzed using a machine that is connected to the canopy/hood.

Participants will be discharged from the hospital, and research staff will escort them to the Center for Weight and Eating Disorders where their body composition will be measured using dual energy X-ray absorptiometry (DEXA). During this test, X-ray pictures of their body will measure how much fat and muscle are present. They will lie flat on a table and a machine will take pictures of different areas of the body. This test will last about 30 minutes. This will conclude the assessment visit.

Eating Conditions & Assessments Upon completion of the baseline assessment, participants will be randomly assigned to start with one of two eating conditions: 1) Daytime or 2) Delayed, and then they will switch and eat on the other schedule for the final part of the study. If they are assigned to the Daytime eating condition first, they will be asked to consume all of their meals and snacks each day between 8 am and 7 pm. If they are assigned to the Delayed eating condition first, they will be asked to consume all of their meals and snacks between 12 pm and 11 pm each day. They will eat on these schedules for 8 weeks each.

During the two 8-week eating condition periods, all of their meals and snacks will be provided by the research kitchen and will be delivered to them by a member of the research staff twice per week. They will be provided a personalized menu and asked to track each food item they consume. They will also be asked to record any beverages they consume on this menu (beverages will not be provided). If occasionally they do not eat the meals provided, they will be asked to use their smart phone or electronic device to send a picture of their food to the study team before they eat it, and again if any food is not eaten when they have finished their meal. They will be asked to wear an Actigraph for the duration of the study, and study staff will deliver new devices and collect used devices one time per week. They will be sent and asked to respond to daily queries by text message or email regarding their eating, sleeping, and exercise. At the end of the 8 weeks, they will complete the second overnight assessment visit (as described above).

For two weeks following this second assessment, they will be asked to eat as they normally would. During this "wash-out" period they will eat what and when then would like. They will then complete the third overnight assessment visit before starting the second eating condition (Delayed for those initially assigned to the Daytime schedule; Daytime for those initially assigned to the Delayed schedule). They will be asked to eat on this new schedule for 8 weeks. They will then complete the fourth and final overnight assessment. After this final assessment visit, their participation in the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Adults of all races and ethnicities
* Age 21-45; BMI 20-27 kg/m2
* stable weight (+/- 10 lbs) over the previous 6 months
* Women must be pre-menopausal with regular menstrual cycles.

Exclusion Criteria:

* Regular exercise more than 3 d/wk, for 30 min measured by exercise logs and actigraphy
* normal activity levels are required throughout the study (+/-30 min/wk of baseline level).
* Unstable, serious medical conditions
* use of medicine linked to weight gain/loss
* cancer, diabetes, or autoimmune disease
* use of illicit drugs, melatonin, diuretics or hypnotics
* current weight loss program; presence of a sleep disorder (determined by surveys and actigraphy)
* night shift work; extreme chronotypes (extreme larks or night owls)
* habitual waking outside of 0600 h-0930h
* habitual bedtime outside of 2200h to 2400h
* sleep duration outside of 6.5 to 8.5 h/night.
* Psychiatric exclusions will be depression (Patient Health Questionnaire-9 score 9), lifetime bipolar disorder, psychosis, or lifetime eating disorder; or any other severe psychiatric disorder judged to interfere with study adherence as assessed by the Structured Clinical Interview for the DSM-IV.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, PhD, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Center for Weight and Eating Disorders, Perelman School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allison KC, Hopkins CM, Ruggieri M, Spaeth AM, Ahima RS, Zhang Z, Taylor DM, Goel N. Prolonged, Controlled Daytime versus Delayed Eating Impacts Weight and Metabolism. Curr Biol. 2021 Feb 8;31(3):650-657.e3. doi: 10.1016/j.cub.2020.10.092. Epub 2020 Nov 30. PMID 33259790

RESULTS

PARTICIPANT FLOW:
Groups:
- Daytime Condition (8 Wks), Followed by Washout (2 Wks), Followed by Delayed Condition (8 Wks): Participants were asked to eat on the Daytime condition first, eating all of their meals and snacks, as provided by the study, between 0800 and 1900 hr for 8 weeks. They then had a 2-week washout period eating as they liked. Finally, they were on the Delayed condition when they ate their meals between 1200 and 2300 hr for 8 weeks.
- Delayed Condition (8 Wks), Followed by Washout (2 Wks), Followed by Daytime Condition (8 Wks): Participants were asked to eat on the Delayed condition first when they ate their meals between 1200 and 2300 hr for 8 weeks. They then had a 2-week washout period eating as they liked. Finally, they were on the Daytime condition, eating all of their meals and snacks, as provided by the study, between 0800 and 1900 hr for 8 weeks.
Period: Overall Study
Arm/Group | Daytime Condition (8 Wks), Followed by Washout (2 Wks), Followed by Delayed Condition (8 Wks) | Delayed Condition (8 Wks), Followed by Washout (2 Wks), Followed by Daytime Condition (8 Wks)
Started | 9 | 8
Completed | 7 | 5
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: All participants complete all of the eating conditions and washout period, so they are included as one group in the baseline analysis population.
Groups:
- All Study Participants: Participants will be asked to eat all of their meals and snacks, as provided by the study, between 0800 and 1900 during the Daytime condition and between 1200 to 2300h in the Delayed condition.
  Participants will be randomly assigned to eat per the prescribed eating condition for 8 weeks during eating condition 1. They will then have a 2-week washout period. They will complete the alternate eating condition for 8 weeks during eating condition 2.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 3
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 1
  Race: White | 13
  Race: More than one race | 0
  Race: Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 65.10 (7.09)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Changes Between the Daytime vs. Delayed Eating Conditions
Description: To determine if timing of food consumption (daytime vs. delayed eating) affects body mass (kg).
Time Frame: pre-post changes between the daytime and delayed eating conditions; change for each condition is calculated from measures at baseline and 8 weeks (end of condition)
Population: All participants completed both eating conditions in a cross-over design and are included in the analyses for the outcomes for each eating condition.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Daytime Eating Condition: Eating Condition: Participants will be randomly assigned to eat between 8 am and 7 pm for 8 weeks
- Delayed Eating Condition: Eating Condition: Participants will be randomly assigned to eat between 12 pm and 11 pm for 8 weeks.
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 12 | 12
kg | -1.1 (1.6) | 0.2 (1.3)

2. Secondary Outcome: Respiratory Quotient Changes in the Daytime vs Delayed Eating Conditions
Description: Changes in fuel oxidation as measured by respiratory quotient with indirect calorimetry.
Time Frame: as for outcome 1
Population: All participants were analyzed together for each outcome measure in this crossover study as all participants completed each eating condition.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 12 | 12
unitless | -.012 (.038) | -.021 (.062)

3. Secondary Outcome: Energy Expenditure Changes Between the Daytime and Delayed Eating Conditions
Description: Changes in resting energy expenditure as measured by indirect calorimetry before and after each eating condition.
Time Frame: as for outcome 1
Population: All participants were analyzed in for both eating conditions as this was a crossover study where participants completed both eating conditions.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Daytime Eating Condition | Delayed Eating Condition
Number analyzed (Participants) | 12 | 12
kcal/day | -93.66 (97.74) | 24.35 (182.90)

ADVERSE EVENTS:
Time Frame: approximately 18 weeks
Description: We collected adverse event information across each of the two eating conditions (8 weeks each) and the washout period (2 weeks), for a total of approximately 18 weeks for each participant across the 2 years and 7 months of the trial when participants were active. This time varied in case of study drop out or scheduling issues that may have impacted the exact length of the washout or eating conditions.
Groups:
- Daytime Eating Condition Followed by 2 Week Washout, Followed by Delayed Eating Condition: Participants will be asked to eat all of their meals and snacks, as provided by the study, between 0800 and 1900 followed by a 2 week washout, followed by eating on the delayed condition (1200 to 1900) for eight weeks.
- Delayed Eating Condition Followed by 2 Week Washout, Followed by Daytime Eating Condition: Participants will be asked to eat all of their meals and snacks, as provided by the study, between 1200 and 2300 followed by a 2-week washout, followed by eating on the daytime condition (0800 to 1900) for eight weeks.
Arm/Group | Daytime Eating Condition Followed by 2 Week Washout, Followed by Delayed Eating Condition | Delayed Eating Condition Followed by 2 Week Washout, Followed by Daytime Eating Condition
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04414644/Prot_SAP_001.pdf
  • Informed Consent Form (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04414644/ICF_000.pdf